CLINICAL TRIAL: NCT00526305
Title: LAL-Ph-2000: Treatment of Acute Lymphoblastic Leukemia Chromosome Philadelphia Positive
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: PETHEMA Foundation (Other)
Responsible Party: Pethema, pethema
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LAL-Ph-2000
Record Dates: First submitted 2007-09-05; First posted 2007-09-10 (Estimated); Last update posted 2010-01-05 (Estimated); Status verified 2010-01

CONDITIONS: Acute Lymphoblastic Leukemia
Keywords: Acute Lymphoblastic Leukemia; Chromosome Philadelphia positive
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Vincristine; Daunorubicin; Prednisone; Asparaginase; Mitoxantrone; Cytarabine; Hydrocortisone; Mercaptopurine; Cyclophosphamide; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Vincristine — 1,5 mg/m2 i.v., days 1 and 8
Drug: Daunorubicin — 60 mg/m2, i.v., days 1 and 8
Drug: Prednisone — 60 mg/m2 day, i.v. or oral, days 1 to 14
Drug: L-Asparaginase — 10.000 UI/m2, i.v., days 5-7 and 11-13. Total: 6 doses.
Drug: Mitoxantrone — 12 mg/m2 i.v days 15, 16 and 17
Drug: Cytosine Arabinoside — 1.500 mg/m2 /12 hours, days 16, 17 and 18 (total: 6 doses) If slow response to treatment: 3.000 mg/m2/12 hours, days 18, 19, 20 and 21 (8 doses)
Drug: Hydrocortisone — 10 mg ,15 mg or 20 mg depending of age
Drug: Mercaptopurine — 50 mg/m2, oral, days 1 to 7, 28-35 and 56-63 in consolidation
Drug: Cyclophosphamide — 600 mg/m2 day, i.v., days 1 to 15 in consolidation
Drug: Dexamethasone — 10 mg/m2 day, oral or i.v. days 1-14 5 mg/m2 day, oral. or i.v., days 15-21

SUMMARY:
Due to ALL Ph+ patients should receive a different treatment, is proposed a therapeutical protocol with: intensification treatment of induction to increment the CR rate, allogenic transplantation in first CR, autologous transplantation follow by alfa interferon in patients cannot done allogenic transplantation.

DETAILED DESCRIPTION:
Remission Induction:

* Vincristine (VCR): 1,5 mg/m2 i.v., days 1 and 8
* Daunorubicin (DNR): 60 mg/m2 i.v., days 1 and 8.
* Prednisone (PDN): 60 mg/m2/day, i.v. or p.o., days 1 to 14
* L-asparaginase (L-ASA): 10.000 UI/m2, i.v.days 5-7 and 11-13

Results:

1. Standard response: The induction treatment will be completed with the same drugs, changing L-ASA to ARA-C, during two more weeks

2 Slow response. Chemotherapy with mitoxantrone and high dose ARA-C

Intrathecal chemotherapy:

Treatment with mitoxantrone, ARA-C e hydrocortisone, days 1 and 22

CONSOLIDATION TREATMENT 1

Start in two weeks after last dose of induction chemotherapy:

* Mercaptopurine (MP) 50 mg/m2, p.o., days 1-7, 28-35 and 56-63
* Mitoxantrone (MTX): 3g/m2, i.v., in 24 hours, day 1, 28 and 56.
* VM-26: 150 mg/m2 every 12 horas, i.v. (infusión 1 hora), días 14 y 42
* ARA-C: 500 mg/m2 cada 12 hours, i.v., in 3 hours, days 14-15 and 42-43
* Intrathecal treatment, days 28 and 56.

6.4. CONSOLIDATION TREATMENT 2

Start in a week after last dose of mercaptopurine of previous cycle

* Dexamethasone (DXM):
* 10 mg/m2 day, p.o. or i.v. days 1-14
* 5 mg/m2 day, p.o. or i.v., days 15-21
* Vincristine (VCR): 1,5 mg/m2 i.v., days 1 and 8 and 15
* Daunorubicin (DNR): 30 mg/m2 i.v., days 1, 2, 8 and 9.
* CFM 600 mg/m2 day, i.v., days 1 and 15
* L-asparaginase (L-ASA): 10.000 UI/m2, i.v.or im , days 1-3 and 15-17
* Intrathecal treatment days 1 and 15.

TRANSPLANTATION

Hematopoietic autologous transplantation with related donor, one or two months after last dose of consolidation treatment.

Hematopoietic autologous transplantation with unrelated donor, in patients younger than 45, and with PS 0-1

Hematopoietic autologous transplantation in patients without related donor and without unrelated donor after six months searching

ELIGIBILITY:
Inclusion Criteria:

ALL BCR/ABL+ patients Age < 65 years No previous treatment

Exclusion Criteria:

1. Other LLA variability
2. Previous history of coronary valvular, hypertensive cardiopathy illness
3. Chronic hepatic illness
4. Chronic respiratory insufficiency
5. Renal insufficiency not caused by LLA
6. Severe neurological problems not caused by LLA
7. Severe affection of the performance status (grade 3-4 OMS gradation) not caused by LLA

Max Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2000-01; Primary Completion 2005-04 (Actual); Study Completion 2005-04 (Actual)

PRIMARY OUTCOMES:
To evaluate the efficacy of treatment in order to response rate, relapse free survival and overall survival | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Ribera Josep Mª, Dr, Study Chair — Germans Trias i Pujol Hospital
Locations (50):
- Spain (50):
  - Hospital General de Alicante, Alicante, Alicante
  - Hospital Ntra. Sra. Sonsoles, Ávila, Avila
  - Hospital Clínic, Barcelona, Barcelona
  - Hospital del Mar, Barcelona, Barcelona
  - Hospital vall d'Hebrón, Barcelona, Barcelona
  - Hospital general de Castellón, Castelló, Castellón
  - Hospital Arnau de Vilanova, Lleida, Lleida
  - Hospital Clínico San Carlos de Madrid, Madrid, Madrid
  - Hospital General Universitario Gregorio Marañón, Madrid, Madrid, Madrid
  - Hospital Universitario de la Princesa, Madrid, Madrid
  - Hospital General Universitario Morales Meseguer., Murcia, Murcia
  - . Hospital Clínico Universitario Virgen de la Victoria, Málaga, Málaga
  - Hospital de Navarra, Pamplona, Navarre
  - Hospital Central de Asturias, Oviedo, Principality of Asturias
  - Hospital Verge de la Cinta, Tortosa, Tarragona
  - Hospital Clínico Universitario de Valencia, Valencia, Valencia
  - Hospital Clínic, Valencia, Valencia
  - Hospital dr. Peset, Valencia, Valencia
  - Hospital General Universitario, Valencia, Valencia
  - Hospital La Fe, Valencia, Valencia
  - Hospital Clínico Lozano Blesa, Zaragoza, Zaragoza
  - Complejo Hospitalario Universitario de Albacete, Albacete
  - Hospital de Badalona Germans Trias i Pujol, Badalona
  - Hospital de Sant Pau, Barcelona
  - Basurtuko Ospitalea, Basurto
  - Hospital de Cruces, Bilbao
  - Hospital de Jerez de la Frontera, Jerez de la Frontera
  - Complejo Hospitalario León, León
  - Complexo Hospitalario Xeral-Calde, Lugo
  - Clínica Puerta de Hierro, Madrid
  - Hospital 12 de Octubre, Madrid
  - Hospital de la Princesa, Madrid
  - Althaia, Xarxa Asistencial de Manresa, Manresa
  - H. Carlos Haya, Málaga
  - Hospital General Morales Meseguer, Murcia
  - Hospital Santa María del Rosell, Murcia
  - Complejo Asistencial Son Dureta, Palma de Mallorca
  - Hospital Son Llatzer, Palma de Mallorca
  - Clínica Universitaria de Navarra, Pamplona
  - Complejo Hospitalario de Pontevedra_Hospital Montecelo, Pontevedra
  - Corporació Sanitaria Parc Taulí, Sabadell
  - Hospital de Sagunto, Sagunto
  - Hospital Clínico Universitario de Salamanca, Salamanca
  - Hospital Universitario de Canarias, Santa Cruz de Tenerife
  - Complejo Hospitalario Universitario de Santiago, Santiago de Compostela
  - Hospital General de Segovia, Segovia
  - H.U. Virgen del Rocio, Seville
  - Hospital Clínico de Valladolid, Valladolid
  - Complejo Hospitalario Universitario de Vigo, Vigo
  - Hospital de Galdakao, Vizcaya

REFERENCES:
- See also: Spanish Association of Haematology — http://www.aehh.org